CLINICAL TRIAL: NCT02735746
Title: Novel High Fidelity Functional Lung Imaging in Adults Undergoing Radiation Therapy to Assess for Radiation Pneumonitis
Brief Title: Novel Lung Imaging in Adults Undergoing Radiation Therapy to Assess for Radiation Pneumonitis
Acronym: HFFLI
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Shiao, Assistant Professor, Cedars-Sinai Medical Center
Other Study IDs: IIT2015-07-SHIAO-HIFIDELI
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Breast Cancer; Mediastinum Lesion; Radiation Pneumonitis
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Radiation Pneumonitis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- High fidelity functional lung imaging: High fidelity functional lung imaging (HFFLI) is an improved method of measuring pulmonary function by analyzing 3-Dimensional (3D) motion. Using this technique, we are able to detect and localize pathological changes in the lung with sub-segmental resolution. The approach uses a unique cross-correlation analysis and non-linear optimization to reconstruct lung tissue motion from a small number of standard projections. All participants will undergo standard 4D Computed Tomography (CT), standard Cone Beam CT, research Low-dose Cinefluorography, and additional research Pulmonary Function Tests.
  Interventions: Radiation: 4D Computed Tomography (CT); Radiation: Cone Beam CT; Radiation: Low-dose Cinefluorography; Device: Pulmonary Function Tests

INTERVENTIONS:
Radiation: 4D Computed Tomography (CT) — The initial 4DCT imaging obtained as part of a subject's planning CT for their standard radiation treatment.
Radiation: Cone Beam CT — Daily cone beam CT imaging at each radiation treatment visit, as part of standard care
Radiation: Low-dose Cinefluorography — A series of images consisting of five six-second cinefluorographs (real time fluoroscopic movies, for a total each time of 30 seconds of fluoroscopy) of the lungs while the subject is breathing, each at precisely measured angles to the subject, on 4 different occasions.
  Other Names: Fluoroscopic images
Device: Pulmonary Function Tests — Pulmonary Function Testing (PFT) gives global functional data for the lungs as a whole, but is relatively insensitive to early pathological changes. It involves taking very deep breaths and exhaling as forcefully as possible.
  Research PFTs will be conducted at 4 and 12-months post radiation therapy

SUMMARY:
The purpose of this study is to to compare lung function data generated by applying High Fidelity Functional Lung Imaging (HFFLI) software to 4D CT, cone beam CT, and fluoroscopic images of the lungs breathing to determine whether different modalities of imaging provide similar data on lung movement and function. HFFLI may detect changes in lung function in patients undergoing External Beam Radiotherapy for cancer.

DETAILED DESCRIPTION:
This study is designed to test a novel technology to examine early changes in the lung in hopes of identifying patients who may be at risk for radiation pneumonitis. Eligible subjects will undergo standard of care treatment with the use of the Varian TrueBeam system for radiation therapy of a cancer lesion in the chest. The imaging data acquired as part of usual standard of care for these patients is a pre-treatment 4D planning CT scan, and a daily cone beam CT at each radiation treatment visit. We will also obtain a series of images consisting of five six-second cinefluorographs (real time fluoroscopic movies, for a total each time of 30 seconds of fluoroscopy) of the lungs while the subject is breathing, each at precisely measured angles to the subject, on 4 different occasions. This study will compare lung function data generated by applying High Fidelity Functional Lung Imaging (HFFLI) software to 4D CT, cone beam CT, and fluoroscopic images of the lungs breathing to determine the degree of correlation between data generated from different imaging modalities. The study is open to adults over the age of 18, at any stage of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Prospective subjects will have been referred to Radiation Oncology for treatment requiring the use of the Varian TrueBeam system, for radiation therapy of a cancer lesion in the chest wall, lung, breast, or mediastinum in which the radiation field will include a portion of lung
* The subject is able to understand the risks, benefits, and possible alternatives to participation in the study, and is able to give both written and verbal voluntary informed consent

Exclusion Criteria:

* For any reason, including pregnancy, subject is considered by the Investigator to be an unsuitable candidate or is put at excess risk by the study procedures.
* Significant existing lung disease, not related to cancer as determined by the PI's review of the patient's PFTs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18, referred to Radiation Oncology for treatment requiring the use of the Varian TrueBeam system for radiation therapy of a cancer lesion in the chest.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-08-21 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
A Pearson correlation of >0.579 between peak expiratory flow as measured by HFFLI analysis of cinefluorograph compared with 4D planning CT | Baseline
A Pearson correlation of >0.579 between peak inspiratory flow as measured by HFFLI analysis of cinefluorograph compared with 4D planning CT | Baseline
A Pearson correlation of >0.579 between ventilation/local time constant as measured by HFFLI analysis of cinefluorograph compared with 4D planning CT | Baseline
A Pearson correlation of >0.579 between expiratory time constant as measured by HFFLI analysis of cinefluorograph compared with 4D planning CT | Baseline
A Pearson correlation of >0.579 between inspiratory time constant as measured by HFFLI analysis of cinefluorograph compared with 4D planning CT | Baseline
A Pearson correlation of >0.579 between tissue shear as measured by HFFLI analysis of cinefluorograph compared with 4D planning CT | Baseline
A Pearson correlation of >0.579 between peak expiratory flow as measured by HFFLI analysis of cinefluorograph compared with cone beam CT | During radiation therapy
  As part of standard care, patients will have a cone beam CT on each day they receive radiation treatment. Treatment period varies.
A Pearson correlation of >0.579 between peak inspiratory flow as measured by HFFLI analysis of cinefluorograph compared with cone beam CT | During radiation therapy
  As part of standard care, patients will have a cone beam CT on each day they receive radiation treatment. Treatment period varies.
A Pearson correlation of >0.579 between ventilation/local time constant as measured by HFFLI analysis of cinefluorograph compared with cone beam CT | During radiation therapy
  As part of standard care, patients will have a cone beam CT on each day they receive radiation treatment. Treatment period varies.
A Pearson correlation of >0.579 between expiratory time constant as measured by HFFLI analysis of cinefluorograph compared with cone beam CT | During radiation therapy
  As part of standard care, patients will have a cone beam CT on each day they receive radiation treatment. Treatment period varies.
A Pearson correlation of >0.579 between inspiratory time constant as measured by HFFLI analysis of cinefluorograph compared with cone beam CT | During radiation therapy
  As part of standard care, patients will have a cone beam CT on each day they receive radiation treatment. Treatment period varies.
A Pearson correlation of >0.579 between tissue shear as measured by HFFLI analysis of cinefluorograph compared with cone beam CT | During radiation therapy
  As part of standard care, patients will have a cone beam CT on each day they receive radiation treatment. Treatment period varies.

SECONDARY OUTCOMES:
Forced expiratory volume 1 (FEV1) | At 12 months post radiation
FEV1/Forced vital capacity | At 12 months post radiation
Total lung capacity | At 12 months post radiation
Diffusing capacity for carbon monoxide | At 12 months post radiation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shiao, MD, PhD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No